CLINICAL TRIAL: NCT06539520
Title: Impact of Aerobic Training on Cardio-respiratory Fitness and Health Related Quality of Life in Stroke Survivors
Brief Title: Aerobic Training on Cardio-respiratory Fitness and Health Related Quality of Life
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Adly A Adam (Other)
Responsible Party: Sponsor-Investigator, Adly A Adam, Lecturer Physical Therapy, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P.T.REC/012/003588
Record Dates: First submitted 2024-07-29; First posted 2024-08-06 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Hemiplegia, Spastic
MeSH Terms: conditions — Hemiplegia

STUDY DESIGN:
Intervention Model Description: Prospective, pre-posttreatment, randomized controlled trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Another researcher via an opaque envelopes involved number defining the 80 post stroke participants, then randomly allocated.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic Training Group A (Experimental): Forty post-stroke patients will receive aerobic training program, plus selected physical therapy program.
  Interventions: Other: Aerobic training program; Other: Selected physical therapy program for post stroke patients
- Control Group B (Other): Forty post-stroke patients will receive selected physical therapy program.
  Interventions: Other: Selected physical therapy program for post stroke patients

INTERVENTIONS:
Other: Aerobic training program — Aerobic training program; on interval moderate mode, 3 session per week, for 16 weeks, along 30-40 minutes, plus 5-10 minutes of warm up and 5 minutes cooling down, with 50-80% of maximal heart rate for each patient based on age. that progress every month by 10% directed by rating of perceived exertion.
  Arms: Aerobic Training Group A
Other: Selected physical therapy program for post stroke patients — Selected neurorehabilitation for 1 hour session; 3 sessions per week, for 16 weeks. It involves weight shift side to side, reaching toward weak side, shoulder flexion overhead, shoulder external rotation, overhead press, shoulder internal rotation with Thera-band, heel slides, bridging, lying terminal knee extension, toe and heel raises, sensory reeducation exercises, and body awareness therapy.

SUMMARY:
Stroke is a major health problem among Egyptian population; an obvious raise in stroke prevalence in all Egyptian governorates. Most stroke survivors commonly develop disabilities those were correlated with restricted physical activity levels. Stroke survivors' cardio-respiratory fitness has several negative impacts such as elevated risk of being affected by other cardiovascular diseases. So, the current study will be conducted to cover the lack in literature concerning the effect of aerobic training on cardiovascular endurance in stroke survivors aiming to faster recovery and reduce the risk of cardiac dysfunction and recurrent strokes.

DETAILED DESCRIPTION:
Stroke as a cerebrovascular accident has a significant prevalence, as well it was addressed a one of major etiologies for other comorbidities, even mortality. Where, cardiac rehabilitation is a structured exercise program that almost designed to offer an opportunity to break the inactivity cycle, reduce associated cardiovascular risks, also improve perceived confidence and quality of life in stroke survivors . Therefore, aerobic training could be defined as a core component that focuses on cardio-respiratory fitness, walking speed and endurance for stroke survivors. Up on that, this clinical trial will be conducted to investigate the effect of aerobic training on cardiorespiratory fitness and health related quality of life in stroke survivors. It will be conducted on eighty post stroke patient (hemiplegic; 55-65 years old with functional ambulatory category more than 3) from Outpatient clinic of neurological department of El-Kasr El-Aini Hospital. They will be allocated into 2 groups; Group A will involves 40 patients will receive aerobic training program, plus traditional physical therapy program. While, Group B will involves 40 patients will receive traditional physical therapy program only. 6-Menutes walk test, Stroke impact scale are the outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Both genders,
* Age range is 55-65 years old,
* Within one year post ischemic stroke,
* Right or left sided stroke,
* hemiplegic and hemiparetic patients,
* Medications include anti-spastics, Beta blockers, ACE inhibitors, and diuretics.
* Functional ambulatory category of three or more,
* Hemodynamic stable,
* Did not participate in any other research study within at least 3 months.

Exclusion Criteria:

* Sever anemia,
* Uncontrolled hypertension, or diabetes mellitus,
* Recent cardiothoracic surgeries,
* Cognitive disorders 'mini mental state exam less than 24'
* Auditory and visual problems,
* Dementia,
* Modified Rankin score 3 or more,
* Seizure,
* Musculoskeletal disorders,
* Stroke or serious head trauma within last 3 months,
* Vertrobrobasilar stroke,

Ages: 55 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
6-Minutes walk test | Baseline of the study, and after 16 weeks at the end of the study.
  A sub-maximal exercise test will be used to assess aerobic capacity and endurance, and functional capability of stroke survivors. 6-Minutes walk test requires stop watch, measuring/ trundle wheel, 30 meter stretch of unimpeded walk way, 2 cones, pulse oximeter, and Borg breathlessness scale. It has excellent reliability, validity, and responsiveness. Its' gained scoring values will be expressed in meters that if more indicates better recovery.

SECONDARY OUTCOMES:
Stroke Impact Scale | Baseline of the study, and after 16 weeks at the end of the study.
  A stroke-specific, self-reported, health status measure. It is designed to assess multi-dimensional stroke outcomes involving strength (4 items), hand function (5 items), activities of daily living/ instrumental activities of daily living (10 items), mobility (9 items), communication (7 items), emotion (9 items), memory (7 items), and participation (8 items). The over score ranged from Zero indicating no recovery up to 100 indicating full recovery

CONTACTS AND LOCATIONS:
Overall Officials: Ali F Rahmy, PHD, Study Director — Professor of Cardiovascular, Respiratory Disorders
Locations (1):
- El-Tahrir st.- in front of Ben El-Sarayat, Ad Doqi Al Giza, Giza Governate, Giza, Egypt